CLINICAL TRIAL: NCT06320912
Title: A Prospective, Multicenter, Randomized Controlled, Non-inferiority Clinical Study Evaluating the Efficacy and Safety of Intraparenchymal Portal Vein Covered Stents for the Treatment of Portal Hypertension and Its Complications
Brief Title: Efficacy and Safety of Intraparenchymal Portal Vein Covered Stents in Treating Portal Hypertension and Its Complications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Shenqi Medical Technology Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TIPS01
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-01

CONDITIONS: Portal Hypertension
Keywords: Portal hypertension
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group(A) (Experimental)
  Interventions: Device: The intraparenchymal portal vein covered stent
- Group(B) (Active Comparator)
  Interventions: Device: TIPS Covered Stent System GORE

INTERVENTIONS:
Device: The intraparenchymal portal vein covered stent — The intraparenchymal portal vein covered stent, produced by Shanghai Shenqi Medical Technology Co., Ltd., is used for a transjugular approach. It establishes an artificial shunt between the hepatic vein and the main branches of the portal vein within the liver. This helps in reducing portal venous pressure and alleviating or improving the symptoms of portal hypertension and its complications, such as variceal bleeding, gastropathy, refractory ascites, and/or hepatic hydrothorax.
  Arms: Group(A)
Device: TIPS Covered Stent System GORE — The GORE® VIATORR® Transjugular Intrahepatic Portosystemic Shunt (TIPS) Covered Stent consists of an implantable covered stent and a percutaneous delivery catheter.
  Arms: Group(B)

SUMMARY:
The objective of this study is to assess the non-inferiority of the intraparenchymal portal vein covered stent in terms of safety and efficacy for managing portal hypertension and its related complications, in comparison to the currently available TIPS Covered Stent System by GORE.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized controlled, non-inferiority clinical trial. It plans to enroll approximately 258 qualified participants from about 25 research centers nationwide. Participants will be randomly assigned in a 1:1 ratio to either the experimental group or the control group for the treatment of portal hypertension and its related complications. The primary endpoint of the study is the patency rate of the stents 12 months after the initial surgery. All participants will undergo clinical follow-ups at 1 month, 6 months, and 1 year post-stent implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years (inclusive); male or non-pregnant female.
* Diagnosed with cirrhosis and associated complications of portal hypertension (such as esophageal and gastric variceal bleeding, refractory ascites), and meeting the consensus recommendations for TIPS indications (see Appendix 5).
* Participants must understand the purpose of the trial, voluntarily participate, sign an informed consent form, and be willing to complete the follow-up according to the project requirements.

Exclusion Criteria:

* Severe right heart failure, congestive heart failure (LVEF < 40%), or severe valvular heart dysfunction.
* Uncontrolled systemic infection or inflammation.
* Persistent moderate to severe pulmonary hypertension after treatment (tricuspid regurgitant peak velocity > 3.4 m/s or pulmonary artery systolic pressure > 50 mmHg).
* Patients in hepatic encephalopathy coma or comatose phase (West Haven Criteria Stage III, IV).
* Severe liver dysfunction, Child-Pugh score > 13, or MELD score > 18.
* Serum creatinine (Scr) > 178 umol/L or on dialysis.
* Stage IIIa or higher liver malignancy.
* Budd-Chiari syndrome, hepatic veno-occlusive disease, or obstructive cholestasis.
* Polycystic liver disease.
* Unrectifiable coagulopathy (INR > 5 or PLT count < 20 x 10^9/L).
* Main portal vein thrombosis occupying > 50% of the lumen area or cavernous transformation of the portal vein.
* Previous TIPS procedure or planned liver transplantation within a year.
* Allergy to contrast agents or nickel-titanium alloys.
* Life expectancy less than 1 year.
* Participation in other drug or medical device clinical trials within three months before screening.
* Other conditions deemed by the researcher as unsuitable for participation in this clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2024-04-05 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative Stent Patency Rate | 12 months
  In the absence of a secondary intervention, portal venography indicates a luminal narrowing of ≤50% and a portal pressure gradient (PPG) of ≤12mmHg or a reduction of ≥50% from the baseline value prior to the surgery.

SECONDARY OUTCOMES:
Immediate Postoperative Technical Success Rate | Immediate postoperative
  Successful insertion and smooth withdrawal of the covered stent and delivery system, successful establishment of a shunt, accurate positioning of the stent, and postoperative angiography showing ≤30% diameter narrowing.
Incidence of Secondary Interventions at 1 Month, 6 Months, and 12 Months Postoperatively | 1 Month, 6 Months, and 12 Months
Incidence of Stent Dysfunction at 1 Month, 6 Months, and 12 Months Postoperatively | 1 Month, 6 Months, and 12 Months
Incidence of Major Adverse Events (MAE) at 1 Month, 6 Months, and 12 Months Postoperatively | 1 Month, 6 Months, and 12 Months
All-Cause Mortality Rates at 1 Month, 6 Months, and 12 Months Postoperatively | 1 Month, 6 Months, and 12 Months
Incidence of Grade II or Higher Hepatic Encephalopathy at 1 Month, 6 Months, and 12 Months Postoperatively | 1 Month, 6 Months, and 12 Months
Incidence of Portal Hypertension Rebleeding Confirmed by Endoscopy or Clinical Investigator at 1 Month, 6 Months, and 12 Months Postoperatively (For Original Bleeding Subjects Only) | 1 Month, 6 Months, and 12 Months
Incidence of Ultrasound-Confirmed Recurrence of Grade 2 or Higher Ascites due to Portal Hypertension at 1 Month, 6 Months, and 12 Months Postoperatively (For Subjects with Original Ascites Only) | 1 Month, 6 Months, and 12 Months
Incidence of Adverse Events/Serious Adverse Events | 12 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Medical University Nanfang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No